CLINICAL TRIAL: NCT04645901
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Phase Ia Study in Healthy Adult Subjects to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of SYHA1805
Brief Title: A Study of SYHA1805 in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYHA1805-CSP-001
Record Dates: First submitted 2020-11-17; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYHA1805 (Experimental): Part 1: Subjects will receive a single dose of oral SYHA1805 tablets. Part 2: Subjects will receive single ascending doses of SYHA1805 tablets. Part 3: Subjects will receive a single dose SYHA1805 tablets in a fasted state and a single dose of SYHA1805 tablets after a high-fat, high-calorie meal, with sequence determined by randomization.
  Interventions: Drug: Drug: SYHA1805 tablets
- Placebo (Placebo Comparator): Subjects will receive the matching placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: SYHA1805 tablets — Oral tablets of SYHA1805 with several doses
  Arms: SYHA1805
Drug: Placebo — Oral tablets of placebo with matching several doses
  Arms: Placebo

SUMMARY:
This is a three-part Phase Ia study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses of SYHA1805.

DETAILED DESCRIPTION:
This trial is divided into three parts: 1) The first part: Four Chinese healthy subjects will be included in the pre-test group to evaluate the safety, tolerability and pharmacokinetics after taking SYHA1805 tablets; 2) The second part: To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic characteristics, several single ascending doses of SYHA1805 tablets or matching placebo tablets will be randomly administered to 24 Chinese healthy subjects under fasting condition; 3) The third part :To evaluate the food effect on the pharmacokinetic characteristics, a single dose SYHA1805 tablets will be administered to 12 Chinese healthy subjects under fed or fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 45 years of age inclusive;
* Weight: Body weight ≥50 kg, body mass index (BMI) within the range of 19-28 kg/m2 (inclusive);
* Overtly healthy as determined by medical evaluation including comprehensive physical examinations, vital signs, laboratory examinations, ECG examination, color Doppler ultrasound (abdominal color Doppler ultrasound, heart color Doppler ultrasound), chest X-ray, etc.;
* Agree to use highly effective contraceptive methods (such as condoms or intrauterine devices, contraceptive drugs) during the clinical trial period (screening period to 30 days after the last dose). Male subject refrains from sperm donation;
* Fully understand the content and possible adverse reactions of the test drug, have the ability to communicate with investigators normally, and able to comply with the research requirements(such as: visit on time, and follow the procedures, restrictions and requirements of the protocol);
* Volunteer to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Have history or other underlying risk factors of torsade de pointes ventricular tachycardia, short QT syndrome, long QT syndrome. Have first-degree relatives (biological parents, siblings or children) who suffered from sudden death in young age (less than/equal to 40 years old), drowning or sudden infant death syndrome of unknown cause ;
* Have history of malignant tumors, mental illness, depression, anxiety, and epilepsy;
* Have history of drugs abuse in the past 3 years. or positive drug test at screening;
* Have history of clinically significant drug allergies, or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis), or those who are known to be allergic to experimental drug excipients or the same type of drugs;
* The investigator determines that the subjects have disease that affect drug absorption, distribution, metabolism, or excretion, such as:

  * History of inflammatory bowel disease, gastritis, ulcers, bile duct stones, gastrointestinal or or rectal bleeding;
  * History of major gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, or bowel resection);
  * History or clinical evidence of pancreatic injury or pancreatitis;
  * ALT, AST, and total serum bilirubin are greater than 2 times the upper limits of normal (ULN) or other liver function test abnormalities, and the abnormalities are determined by the investigator to have clinical significance, suggesting liver disease or liver damage;
  * Renal function suggests that the creatinine clearance rate is less than 90 mL/min, or has urinary tract obstruction or difficulty in emptying urine;
* HBsAg positive, HCV-Ab positive, HIV-Ab positive or syphilis antibody positive during the screening period;
* Have history of alcohol abuse within 6 months before screening, have a positive alcohol breath test during the screening period and the baseline period, or cannot stop drinking during the entire study period; Subjects smoke more than 5 cigarettes per day within the 3 months prior to screening, have a positive nicotine test at screening, or cannot give up smoking during the entire study period;
* Have participated in clinical trials of any drug or medical device within 3 months before screening；
* Have undergone major surgery within 3 months before screening, or have had severe infections within 4 weeks before screening;
* Have had significant change in diet or exercise habits within 3 months before screening, such as weight loss, diet, exercise, etc.;
* Donated blood ≥500 mL within 4 weeks before screening, or had severe blood loss in excess of 500 mL, or received blood transfusion within 8 weeks prior to screening;
* Have used any prescription drugs within the 4 weeks before screening, including antibiotics or Chinese herbal medicines; have used any Over-the-Counter (OTC) medications or food supplements (such as vitamins and calcium) within the 2 weeks before screening except for paracetamol (maximum 1000 mg per day), ibuprofen (maximum 2400 mg per day) and topical OTC drugs; have taken a drug within its 5 half-lives prior to the first dose of the study drug;
* Smoking, consumption of alcohol or food/beverages containing xanthine or caffeine, strenuous exercise, or taking foods that affect drug absorption, distribution, metabolism, and excretion (such as grapefruit-containing drinks) within 2 days prior to D-1 ；
* Pregnant or lactating women;
* Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) or non-serious adverse events (AEs) Considered by the Investigator to be Related to Study Drug Administrationorally | Baseline through Day 28
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Baseline through Day 28
  Area under the plasma concentration versus time curve (AUC) after administration of of SYHA1805 under fasting conditions or under the food effect of high-fat, high-calorie meals
Peak Plasma Concentration (Cmax) | Baseline through Day 28
  Peak Plasma Concentration (Cmax) after administration of of SYHA1805 under fasting conditions or under the food effect of high-fat, high-calorie meals
Time to maximum plasma concentration（Tmax） | Baseline through Day 28
  Time to maximum plasma concentration（Tmax）after administration of of SYHA1805 under fasting conditions or under the food effect of high-fat, high-calorie meals
Half time (t1/2) | Baseline through Day 28
  The half time of SYHA1805 after administration are calculated under fasting conditions or under the food effect of high-fat, high-calorie meals
Apparent clearance (CL/F) | Baseline through Day 28
  To assess the apparent clearance (CL/F) after administration of SYHA1805 under fasting conditions or under the food effect of high-fat, high-calorie meals
To evaluate the ECG result of single doses of SYHA1805 administered orally | Baseline through Day 28
  To analysis of the QT Interval after administration of of SYHA1805